CLINICAL TRIAL: NCT01740635
Title: Enhancing Participation In the Community by Improving Wheelchair Skills (EPIC WheelS): A Feasibility Study
Brief Title: EPIC WheelS Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H12-02043
Record Dates: First submitted 2012-11-15; First posted 2012-12-04 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Difficulty Walking
Keywords: rehabilitation; wheelchair; manual wheelchair; wheelchair users; older adults; cognitive computer games; home-based training; community mobility
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPIC WheelS Training Program (Experimental): The EPIC WheelS program includes a comprehensive, structured library of educational material and training activities, organized in a hierarchy from simple to complex. Experimental group subjects will attend 2 training sessions with an expert Trainer. The Trainer will individualize a structured home training program, delivered via a computer tablet, and subjects will train at home for 1 month.
  Interventions: Device: EPIC WheelS Training Program
- Cognitive games (No Intervention): To provide a comparable level of investigator attention, control group subjects will receive two 1-hour social visits. To control for Trainer bias, the experimental and control groups will have separate Trainers. During social visits, the Trainer will discuss subjects' current community activities and their experience using the wheelchair, and provide verbal information related to barriers encountered. Subjects will receive a computer tablet with cognitive stimulation games to account for activity and tablet device exposure. Participants in the extra wheeling sub-group will be instructed to perform additional, unstructured wheeling for 15 minutes, 5 days per week (total 75 minutes/week) and document these on a simple calendar-style form provided. To minimize attrition, control subjects will receive a DVD with a condensed MWC skills education program after the post-intervention data collection is complete.

INTERVENTIONS:
Device: EPIC WheelS Training Program — Subjects will attend an initial assessment/training session and receive a customized home program from their Trainer, which is delivered by way of a portable, interactive computer tablet that can be used for practice in their home or other community venues. After 2 weeks of practice, subjects return for a second 1-hour training session. The Trainer updates their program and they continue practicing at home for another 2 weeks. Subjects will have a caregiver attend all training sessions and supervise their home training. Trainers monitor subject activity remotely and will contact subjects by telephone at the end of weeks 1 and 3 to promote program adherence. Participants in an extra wheeling sub-group will be instructed to perform additional, unstructured wheeling for 15 minutes, 5 days per week and document these on a simple calendar-style form provided.
  Arms: EPIC WheelS Training Program

SUMMARY:
Many older adults have difficulty walking. A wheelchair can improve their participation but older adults typically receive little wheelchair training. Structured training programs are effective but rely on multiple 1:1 sessions with a skilled clinician. EPIC WheelS combines 2 brief training sessions and a 4-week home training program delivered using a portable computer tablet and monitored by an expert trainer. This study investigates the feasibility and potential for using EPIC WheelS with older adult novice wheelchair users in Vancouver and Winnipeg, measuring the impact on wheelchair skill, safety and confidence compared to a control group receiving only cognitive training.

Hypotheses: The investigators expect that the feasibility outcomes will be sufficiently robust to support conducting a subsequent multi-site RCT. The investigators also expect the EPIC WheelS training program will have a significant treatment effect with improvement in wheelchair mobility, compared to a control group.

DETAILED DESCRIPTION:
Many older adults rely on a manual wheelchair (MWC) for community mobility, but are not provided with the skills for independent and effective use of their wheelchair. Suboptimal use of the wheelchair results in substantial social costs such as reduced engagement in meaningful activity, social isolation, and higher caregiver burden. This is a poor use of financial resources, including the cost of wheelchair acquisition and requirements for attendant care. Access to skills training is constrained by the expense and limited availability of skilled therapists; demands of patient and/or clinician travel; and lack of training programs designed specifically for older adults.

Enhancing Participation In the Community by improving Wheelchair Skills (EPIC WheelS) is an individualized home-training program that optimizes learning for older adults while limiting the time demands of expert trainers. Using an affordable mainstream computer tablet device, EPIC WheelS provides a structured training program that can be customized for specific users needs. The tablet is mobile, for in-chair or tabletop use, in home and community locations. A touch screen operated audio-visual display features interactive training and practice activities as well as video-recording capability. Wireless Internet enables user-trainer communication and remote program monitoring and updating by the trainer. A monitored home program that is effective and efficient for older adults has the potential for application to other target groups, particularly those in rural and remote locations with limited access to rehabilitation.

PURPOSE: The purpose is to evaluate the feasibility and effect size estimate of a 1-month customized home training program (EPIC WheelS) for improving wheelchair mobility skills among novice older adult manual wheelchair users compared to usual care. Despite the pervasive use of wheelchairs as an intervention in rehabilitation, the evidence for training in effective wheelchair use is still underdeveloped. Structured training has demonstrated excellent potential, but the most effective and efficient means of providing that training remains unclear. Larger multi-site clinical trials are required to establish evidence to inform and direct clinical practice. The investigators propose that this 2-year feasibility trial is not only critical, but also prudent, prior to moving forward with an expensive large multi-site randomized controlled trial (RCT). Specifically the results of this study will address 1) feasibility outcomes (i.e., recruitment and retention; trainer and subject burden; safety; intervention administration and adherence; perceived benefit) and 2) clinical outcomes (i.e., effect size calculations for the primary and secondary measures). Although the principal intent is feasibility, the sample size calculation is based on the primary clinical outcome to provide a reasonable estimate of an effect size for planning the subsequent large scale RCT.

HYPOTHESES: The investigators expect that the feasibility outcomes will be sufficiently robust to support conducting a subsequent multi-site RCT. The investigators also expect the EPIC WheelS training program will have a significant treatment effect with improvement in wheelchair mobility, compared to a control group. The primary clinical endpoint will be wheelchair skill capacity, as measured by the Wheelchair Skills Test (WST). Secondary clinical outcomes will include wheelchair skill safety; confidence with wheelchair use; mobility; and user evaluation of performance in participation-oriented activities.

ELIGIBILITY:
Inclusion Criteria:

Wheelchair users must

* be at least 50 years old
* use his/her wheelchair for at least 1 hour per day on average
* live within the metropolitan boundaries of Vancouver or Winnipeg
* have a caregiver who is able to attend training sessions and supervise home training

Caregivers must

* be 19 years old or older
* be a caregiver of a manual wheelchair user who is 50 years or older
* able to attend the training sessions
* be able to supervise or spot the wheelchair user during home training

Exclusion Criteria:

Wheelchair users would be excluded if he/she

* cannot communicate or complete the study questionnaires in English
* has a health condition or upcoming procedure that would prevent you from performing training activities (e.g., cancer treatment, surgery)
* is currently receiving wheelchair skills training elsewhere
* cannot use both arms to propel your wheelchair

Caregivers will be excluded if

* he/she cannot communicate in English
* he/she has a health condition or upcoming procedure that would prevent you from supervising training activities (e.g., cancer treatment, surgery)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Wheelchair Skills Test (WST) - Capacity | 4 weeks
  Wheelchair mobility skill capacity will be measured using the Wheelchair Skills Test 4.1 (WST). The WST is a structured assessment with 32 discrete mobility skills required to perform social roles in the community, each scored dichotomously as pass/fail. The WST produces a total Skill Capacity score (0-100%) reflecting the number of skills safely passed. To optimize stability of the measure, increase precision, and control for a learning effect, the WST will be administered twice at baseline and a mean baseline score calculated. Standardized equipment required for the WST (e.g., 5 degree & 10 degree ramps, gravel) is available at both test sites.

SECONDARY OUTCOMES:
Wheelchair Outcome Measure (WhOM) | Baseline, 4 weeks
  The rehabilitation literature strongly suggests that intervention outcomes should include not only externally defined measures, but also measures of user-identified activities of relevance and perceived satisfaction with performance. As part of the baseline data collection, the five most important activities identified with the WhOM will be used to customize the training program for experimental group subjects.
Wheelchair Use Confidence Scale for Manual Wheelchair Users (WheelCon-M 3.0) | Baseline, 4 weeks
  The WheelCon is a self-report questionnaire composed of 65 statements related to confidence using a wheelchair in activities and environments, each rated on a scale from 0 ("not confident") to 100 ("completely confident"), producing a total mean score of 0 - 100.
Life-Space Assessment (LSA) | Baseline, 4 weeks
  The LSA will capture the mobility habits of study subjects. It is a 20-item questionnaire that tracks the locations to which wheelchair users travel on a continuum of 5 environments from the home to outside of town. Subjects report on their movement in each life-space during the past 4 weeks, the frequency of travel, and whether assistance was required.
Health Utility Index 3 | Baseline, 4 weeks
  The Health Utility Index 3 (HUI3) is a brief questionnaire that asks subjects about their health status, reflected in a single-score measure of health-related quality of life (HRQOL).
Wheeling While Talking Test | Baseline, 4 weeks
  The Walking While Talking test will be modified for use with a wheelchair and used to evaluate divided-attention during wheelchair propulsion; we will call this the Wheeling While Talking test.
Wheelchair Skills Test (WST) - Safety | Baseline, 4 weeks
  The WST also provides a total Skill Safety score (0-100%) reflecting the number of skills addressed in a safe manner, regardless of whether the skill is passed or not.
Participant retention rate of 80% | Baseline, 4 weeks
Training adherence (150 minutes/week) rate of 85% | Baseline, 4 weeks
No adverse events reported | Baseline, 4 weeks
Wheeling While Talking test | Baseline, 4 weeks
  Wheelchair mobility is a complex skill and prone to risk for tips, falls and potential injury, particularly with older adult users where motor and cognitive function may decline with age. The Wheeling While Talking test is a new divided-attention assessment for wheelchair users, currently undergoing reliability testing. Collecting data in this study will allow investigation of associations between performance and wheelchair skill, safety and other demographic factors, contributing to validation of this tool.
Data logger | Baseline, 4 weeks
  To capture level of activity while in the wheelchair, a data logger will be mounted on the drive wheel spokes of each participant's wheelchair. The data logger is a small, unobtrusive 'black box' that collects distance and speed via an accelerometer over a period of 6-10 days, depending upon battery life. Collecting this data will allow description and comparison of wheeling patterns and extent of activity among participants. Data loggers will be installed at the first training session and removed at the second training session, approximately 2 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: William C. Miller, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - GF Strong Rehabilitation Centre, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Background] Rushton PW, Miller WC, Mortenson WB, Garden J. Satisfaction with participation using a manual wheelchair among individuals with spinal cord injury. Spinal Cord. 2010 Sep;48(9):691-6. doi: 10.1038/sc.2009.197. Epub 2010 Feb 2. PMID 20125106
- [Derived] Giesbrecht EM, Miller WC. Effect of an mHealth Wheelchair Skills Training Program for Older Adults: A Feasibility Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Nov;100(11):2159-2166. doi: 10.1016/j.apmr.2019.06.010. Epub 2019 Jul 20. PMID 31336101
- [Derived] Giesbrecht EM, Miller WC, Eng JJ, Mitchell IM, Woodgate RL, Goldsmith CH. Feasibility of the Enhancing Participation In the Community by improving Wheelchair Skills (EPIC Wheels) program: study protocol for a randomized controlled trial. Trials. 2013 Oct 24;14:350. doi: 10.1186/1745-6215-14-350. PMID 24156396